CLINICAL TRIAL: NCT02691325
Title: A Single Centre, Three Part, Randomised, Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK2269557 Administered Via the ELLIPTA™ Dry Powder Inhaler to Healthy Subjects
Brief Title: Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK2269557 Administered Via the ELLIPTA Dry Powder Inhaler to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201544
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: ELLIPTA; GSK2269557; Tolerability; Safety; Dry powder Inhaler (DPI); Pharmacokinetics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Charcoal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A (Sequence 1) - Placebo, GSK2269557 200 mcg (Experimental): Subjects will receive a single dose of GSK2269557 matching placebo (one inhalation) in treatment period 1, and single dose of GSK2269557 200 microgram (mcg) (2 inhalations of GSK2269557 100 mcg) in treatment period 2 via the ELLIPTA DPI. The washout period between each dosing day will be at least 14 days. Doses of GSK2269557 may be modified based on emerging data.
  Interventions: Drug: GSK2269557 ELLIPTA DPI; Drug: Placebo ELLIPTA DPI
- Part A (Sequence 2) - GSK2269557 100 mcg, Placebo (Experimental): Subjects will receive a single dose of GSK2269557 100 mcg (one inhalation) in treatment period 1, and single dose of GSK2269557 matching placebo (two inhalations) in treatment period 2 via the ELLIPTA DPI. The washout period between each dosing day will be at least 14 days. Doses of GSK2269557 may be modified based on emerging data.
  Interventions: Drug: GSK2269557 ELLIPTA DPI; Drug: Placebo ELLIPTA DPI
- Part A (Sequence 3) - GSK2269557 100 mcg, GSK2269557 200 mcg (Experimental): Subjects will receive a single dose of GSK2269557 100 mcg (one inhalation) in treatment period 1, and single dose of GSK2269557 200 mcg (2 inhalations of GSK2269557 100 mcg) in treatment period 2 via the ELLIPTA DPI. The washout period between each dosing day will be at least 14 days. Doses of GSK2269557 may be modified based on emerging data.
  Interventions: Drug: GSK2269557 ELLIPTA DPI; Drug: Placebo ELLIPTA DPI
- Part B- GSK2269557 200 mcg (Experimental): Subjects will receive repeated doses of GSK2269557 200 mcg (2 inhalations of GSK2269557 100 mcg) once daily via the ELLIPTA DPI for 10 days. Doses of GSK2269557 may be modified based on emerging data from Part A.
  Interventions: Drug: GSK2269557 ELLIPTA DPI
- Part B- GSK2269557 matching Placebo (Experimental): Subjects will receive repeated doses of GSK2269557 matching Placebo (2 inhalations) once daily via the ELLIPTA DPI for 10 days.
  Interventions: Drug: Placebo ELLIPTA DPI
- Part C- GSK2269557 200 mcg with and without activated charcoal (Experimental): Subjects will receive a single dose of GSK2269557 200 mcg (2 inhalations of GSK2269557 100 mcg) via the ELLIPTA DPI with activated charcoal in one treatment period and without ingestion of activated charcoal in another treatment period. The washout period between each dosing day will be at least 14 days. Dose of GSK2269557 may be modified based on emerging data from Part A.
  Interventions: Drug: GSK2269557 ELLIPTA DPI; Drug: Activated charcoal

INTERVENTIONS:
Drug: GSK2269557 ELLIPTA DPI — GSK2269557 ELLIPTA DPI contains GSK2269557 blended with lactose and magnesium stearate. This will be supplied in two strength of 100 mcg per blister.
  Arms: Part A (Sequence 1) - Placebo, GSK2269557 200 mcg; Part A (Sequence 2) - GSK2269557 100 mcg, Placebo; Part A (Sequence 3) - GSK2269557 100 mcg, GSK2269557 200 mcg; Part B- GSK2269557 200 mcg; Part C- GSK2269557 200 mcg with and without activated charcoal
Drug: Placebo ELLIPTA DPI — Placebo ELLIPTA DPI contains lactose.
  Arms: Part A (Sequence 1) - Placebo, GSK2269557 200 mcg; Part A (Sequence 2) - GSK2269557 100 mcg, Placebo; Part A (Sequence 3) - GSK2269557 100 mcg, GSK2269557 200 mcg; Part B- GSK2269557 matching Placebo
Drug: Activated charcoal — The activated charcoal will be supplied by the clinical site. Charcoal will be administered as a suspension of 5 gram activated charcoal in 40 mL of water. The suspension will be made to drunk, in its entirety.
  Arms: Part C- GSK2269557 200 mcg with and without activated charcoal

SUMMARY:
GSK2269557 is a potent and highly selective inhaled Phosphoinositide 3-Kinase delta inhibitor being developed as an anti-inflammatory and anti-infective agent for the treatment of inflammatory airway diseases. The study will be conducted at a single centre and in 3 Parts. The aim of Part A and B of the study are to assess the safety, tolerability and pharmacokinetics (PK) single and repeat doses of a new formulation of GSK2269557 administered via the ELLIPTA dry powder inhaler (DPI) to healthy subjects. This is the first study in which GSK2269557 will be administered via the ELLIPTA DPI. Part C of the study will investigate the proportion of the systemic exposure that post inhalation is due to the swallowed fraction of the inhaled dose. Part C will also be conducted using the ELLIPTA device and magnesium stearate formulation. Part A will be conducted first. Part B and Part C may be run sequentially or in parallel. Part A is a randomized, double blind, placebo controlled, single dose, dose escalating incomplete block 2-period crossover study in healthy subjects. Subjects will be randomized to receive either one dose strength of GSK2269557 and placebo utilizing placebo replacement, or will receive both active dose strengths. Part B is a randomized, double blind, placebo controlled, repeat dose study in healthy Subjects. Subjects will be randomized to receive either repeat doses of GSK2269557 or placebo for 10 days. Part C is a, randomized, open-label, crossover design to assess the systemic exposure of single doses of GSK2269557 administered via the ELLIPTA DPI to healthy subjects, with and without ingestion of activated charcoal. ELLIPTA is the registered trademark of GlaxoSmithKline groups of companies.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 and 75 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Normal spirometry at Screening (forced expiratory volume in 1 second and forced vital capacity >=80% of predicted - measurements to be taken in triplicate and the highest value must be >=80% of predicted).
* A subject with a clinical abnormality or laboratory parameter(s) outside the reference range for the population being studied may be included only if the investigator, in consultation with the medical monitor if needed, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 18 to 35 kg/square meter (m^2) (inclusive).
* Male subjects. Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until at least 10 days after the last dose of study medication.

  * Vasectomy with documentation of azoospermia.
  * Male condom plus partner use of one of the contraceptive options: Contraceptive subdermal implant, Intrauterine device or intrauterine system, Combined estrogen and progestogen oral contraceptive, Injectable progestogen, Contraceptive vaginal ring and Percutaneous contraceptive patches.
* Female subjects. Female subjects are eligible to participate if they are not pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test at screening and a serum or urine hCG test on admission), not lactating, and at least one of the following conditions applies:

  * Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion , Hysterectomy, Documented Bilateral Oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
  * Female of reproductive potential (FRP) must agrees to the use of male condom with spermicide in addition to one of the following methods from the list of highly effective contraceptive methods from 30 days prior to the first dose of study medication and until at least 10 days after the last dose of study medication: Contraceptive subdermal implant; Intrauterine device or intrauterine system; Combined estrogen and progestogen oral contraceptive; Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches; Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject.

The list does not apply to FRP with same sex partners or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis, when this is their preferred and usual lifestyle. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and protocol.

Exclusion Criteria:

* Asthma or a history of asthma (except in childhood, which has now remitted).
* Alanine Aminotransferase (ALT) and bilirubin >1.5 Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if fractionated and direct bilirubin <35%)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT interval by Fridericia's formula (QTcF) > 450 milliseconds (msec).
* Unable to refrain from the use of prescription drugs (except contraceptives and HRT) or non-prescription drugs (except acetaminophen), including vitamins, herbal and dietary supplements from 7 days before the first dose of study medication until the follow-up visit, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedure or compromise subject safety.
* The subject has received any type of vaccination within 4 weeks of their first dose of study medication, or is expected to be vaccinated within 4 weeks after their last dose of study medication.
* Current smoker or a history of smoking within 6 months of Screening, or a total pack year history of >5 pack years. (number of pack years = [number of cigarettes per day/20] x number of years smoked)
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 alcoholic drinks for males or >7 alcoholic drinks for females. One alcoholic drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 milliliters [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Unable to refrain from the consumption of Seville oranges, grapefruit or grapefruit juice, pummelos, exotic citrus fruits, or grapefruit hybrids from 7 days before all doses of study medication and until collection of the final pharmacokinetic sample in each study period.
* History of sensitivity to any of the study medications, or components thereof (including lactose and Magnesium stearate) or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. Subjects with a positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C Ribonucleic acid (RNA) polymerase chain reaction (PCR) test is obtained.
* A positive test for Human Immunodeficiency Virus(HIV) antibody (according to local policies).
* A positive drug/alcohol screen at screening or on admission (Day -1). - Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* The subject has participated in a clinical trial and has received an investigational product (excluding participation in Part A of this study) within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2016-06-05 (Actual); Study Completion 2016-06-05 (Actual)

PRIMARY OUTCOMES:
Part A: Number of subjects with any adverse event(s) (AE) and serious adverse event(s) (SAE) | Up to 6 weeks
  An AE is any untoward medical occurrence in a clinical investigation subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage.
Part B and C: Number of subjects with any AE and SAE | Up to 4 weeks
  An AE is any untoward medical occurrence in a clinical investigation subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage.
Part A: Systolic and diastolic blood pressure as a measure of safety | Up to 9 weeks
Part B: Systolic and diastolic blood pressure as a measure of safety | Up to 7 weeks
Part C: Systolic and diastolic blood pressure as a measure of safety | Up to 8 weeks
Part A: Heart rate as a measure of safety | Up to 9 weeks
Part B: Heart rate as a measure of safety | Up to 7 weeks
Part C: Heart rate as a measure of safety | Up to 8 weeks
Part A: Temperature as a measure of safety | Up to 9 weeks
Part B: Temperature as a measure of safety | Up to 7 weeks
Part C: Temperature as a measure of safety | Up to 8 weeks
Part A: Respiratory rate as a measure of safety | Up to 9 weeks
Part B: Respiratory rate as a measure of safety | Up to 7 weeks
Part C: Respiratory rate as a measure of safety | Up to 8 weeks
Part A: 12-lead electrocardiogram (ECG) as a measure of safety | Up to 9 weeks
  All scheduled ECGs will be performed after the subject has rested quietly for at least 5 minutes in a supine position.
Part B: 12-lead ECG as a measure of safety | Up to 7 weeks
  All scheduled ECGs will be performed after the subject has rested quietly for at least 5 minutes in a supine position.
Part C: 12-lead ECG as a measure of safety | Up to 8 weeks
Part A: Composite of hematology parameters as a measure of safety | Up to 9 weeks
  The following hematology parameters will be measured: hemoglobin, Hematocrit, Red blood cell (RBC) count, Mean corpuscular volume (MCV), Mean corpuscular hemoglobin (MCH), Platelet count, white blood cell (WBC) count, Total neutrophils (Absolute), Eosinophils (Absolute), Monocytes (Absolute), Basophils (Absolute), and Lymphocytes (Absolute).
Part B: Composite of hematology parameters as a measure of safety | Up to 7 weeks
  The following hematology parameters will be measured: Hemoglobin, Hematocrit, RBC count, MCV, MCH, Platelet count, WBC count, Total neutrophils (Absolute), Eosinophils (Absolute), Monocytes (Absolute), Basophils (Absolute), and Lymphocytes (Absolute).
Part C: Composite of hematology parameters as a measure of safety | Up to 8 weeks
  The following hematology parameters will be measured: Hemoglobin, Hematocrit, RBC count, MCV, MCH, Platelet count, WBC count, Total neutrophils (Absolute), Eosinophils (Absolute), Monocytes (Absolute), Basophils (Absolute), and Lymphocytes (Absolute).
Part A: Composite of chemistry parameters as a measure of safety | Up to 9 weeks
  The following chemistry parameters will be measured: Blood Urea nitrogen (BUN), Uric Acid, Creatinine, Glucose, Calcium, Sodium, Potassium, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Total Bilirubin, Alkaline phosphatase (ALP), Total albumin, Total protein, Total bilirubin and Direct bilirubin.
Part B: Composite of chemistry parameters as a measure of safety | Up to 7 weeks
  The following chemistry parameters will be measured: BUN, Uric Acid, Creatinine, Glucose, Calcium, Sodium, Potassium, AST, ALT, ALP, Total albumin, Total protein, Total bilirubin and Direct bilirubin.
Part C: Composite of chemistry parameters as a measure of safety | Up to 8 weeks
  The following chemistry parameters will be measured: BUN, Uric Acid, Creatinine, Glucose, Calcium, Sodium, Potassium, AST, ALT, ALP, Total albumin, Total protein, Total bilirubin and Direct bilirubin.
Part A: Composite of urinalysis parameters as a measure of safety | Up to 6 weeks
  The following urinalysis parameters will be measured: power of hydrogen (pH), Glucose, Protein, Blood, Ketones by dipstick; specific gravity and Microscopy (if blood or protein is abnormal)
Part B: Composite of urinalysis parameters as a measure of safety | Up to 4 weeks
  The following urinalysis parameters will be measured: pH, Glucose, Protein, Blood, Ketones by dipstick; specific gravity and Microscopy (if blood or protein is abnormal)
Part C: Composite of urinalysis parameters as a measure of safety | Up to 4 weeks
  The following urinalysis parameters will be measured: pH, Glucose, Protein, Blood, Ketones by dipstick; specific gravity and Microscopy (if blood or protein is abnormal)
Part A, B and C: Spirometry measurement as a measure of safety | Screening and Day 1 (Pre-dose and 30 minute (min) post-dose)

SECONDARY OUTCOMES:
Part A and C: Plasma concentrations of GSK2269557 | Pre-dose, 5 min and 30 min, 1 hour (h), 2 h, 4 h, 6 h, 12 h, 24 h post dose of each treatment period
Part B: Plasma concentrations of GSK2269557 | Day 1: pre-dose, and 5 minute (min) and 24 h post-dose (Day 2 pre-dose); Days 6, 7, 8, 9: pre-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h and 24 h post-dose (Day 11), Day 12: 48 h post-dose; and Day 13: 72 h post-dose
Part A and C: Area under the plasma concentration curve (AUC) from time zero to infinity [AUC(0-infinity)] of GSK2269557 following single dose administration | Pre-dose and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h, 12 h, 24 h post dose of each treatment period
Part A and C: AUC from time zero to the time of last quantifiable concentration [AUC(0-t)] of GSK2269557 following single dose administration | Pre-dose and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h, 12 h, 24 h post dose of each treatment period
Part A and C: maximum observed plasma concentration (Cmax) | Pre-dose and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h, 12 h, 24 h post dose of each treatment period
Part A and C: Time to maximum observed concentration (tmax) of GSK2269557 following single dose administration | Pre-dose and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h, 12 h, 24 h post dose of each treatment period
Part A and C: Terminal half life (t1/2) of GSK2269557 following single dose administration | Pre-dose and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h, 12 h, 24 h post dose of each treatment period
Part A and C: concentration at trough (Ctrough) of GSK2269557 following single dose administration | Pre-dose and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h, 12 h, 24 h post dose of each treatment period
Part B: AUC(0-infinity) of GSK2269557 following repeat dose administration | Day 1: pre-dose, and 5 min and 24 h post-dose (Day 2 pre-dose); Days 6, 7, 8, 9: pre-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h and 24 h post-dose (Day 11), Day 12: 48 h post-dose; and Day 13: 72 h post-dose
Part B: AUC(0-t) of GSK2269557 following repeat dose administration | Day 1: pre-dose, and 5 min and 24 h post-dose (Day 2 pre-dose); Days 6, 7, 8, 9: pre-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h and 24 h post-dose (Day 11), Day 12: 48 h post-dose; and Day 13: 72 h post-dose
Part B: Cmax of GSK2269557 following repeat dose administration | Day 1: pre-dose, and 5 min and 24 h post-dose (Day 2 pre-dose); Days 6, 7, 8, 9: pre-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h and 24 h post-dose (Day 11), Day 12: 48 h post-dose; and Day 13: 72 h post-dose
Part B: tmax of GSK2269557 following repeat dose administration | Day 1: pre-dose, and 5 min and 24 h post-dose (Day 2 pre-dose); Days 6, 7, 8, 9: pre-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h and 24 h post-dose (Day 11), Day 12: 48 h post-dose; and Day 13: 72 h post-dose
Part B: t1/2 of GSK2269557 following repeat dose administration | Day 1: pre-dose, and 5 min and 24 h post-dose (Day 2 pre-dose); Days 6, 7, 8, 9: pre-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h and 24 h post-dose (Day 11), Day 12: 48 h post-dose; and Day 13: 72 h post-dose
Part B: Ctrough of GSK2269557 following repeat dose administration | Day 1: pre-dose, and 5 min and 24 h post-dose (Day 2 pre-dose); Days 6, 7, 8, 9: pre-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h and 24 h post-dose (Day 11), Day 12: 48 h post-dose; and Day 13: 72 h post-dose
Part C: AUC from time zero to 24 hours post dose [AUC(0-24)] for GSK2269557 following the inhaled route with and without charcoal | Pre-dose and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h, 12 h, 24 h post dose of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Wilson R, Jarvis E, Montembault M, Hamblin JN, Hessel EM, Cahn A. Safety, Tolerability, and Pharmacokinetics of Single and Repeat Doses of Nemiralisib Administered via the Ellipta Dry Powder Inhaler to Healthy Subjects. Clin Ther. 2018 Aug;40(8):1410-1417. doi: 10.1016/j.clinthera.2018.06.011. Epub 2018 Jul 25. PMID 30055824
- See also: Results for study 201544 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/201544?search=study&b'study_ids=201544'#rs